CLINICAL TRIAL: NCT02810067
Title: Root Coverage With Acellular Dermal Matrix Using the Coronally Positioned Tunnel Technique Comparing Two Different Donor Materials
Brief Title: Root Coverage Comparing an Allograft to a Bovine Xenograft
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was dropped and never started.
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Henry Greenwell, Professor, Director Graduate Periodontics, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17.0534
Record Dates: First submitted 2016-06-20; First posted 2016-06-22 (Estimated); Last update posted 2018-06-18 (Actual); Status verified 2018-06

CONDITIONS: Gingival Recession
MeSH Terms: conditions — Gingival Recession | interventions — Alloderm

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tunnel + AlloDerm® (Active Comparator): A coronally positioned tunnel (CPT) technique for root coverage will be used with acellular dermal matrix (AlloDerm®).
  Interventions: Procedure: Tunnel + AlloDerm
- Tunnel + Novomatrix (Experimental): A coronally positioned tunnel (CPT) technique for root coverage will be used with acellular dermal matrix (Novomatrix).
  Interventions: Procedure: Tunnel + Novomatrix

INTERVENTIONS:
Procedure: Tunnel + AlloDerm — A coronally positioned tunnel (CPT) technique for root coverage will be used with acellular dermal matrix (AlloDerm).
  Other Names: AlloDerm®
  Arms: Tunnel + AlloDerm®
Procedure: Tunnel + Novomatrix — A coronally positioned tunnel (CPT) technique for root coverage will be used with acellular dermal matrix (Novomatrix).
  Other Names: Novomatrix
  Arms: Tunnel + Novomatrix

SUMMARY:
Root coverage with acellular dermal matrix using the coronally positioned tunnel technique comparing two different donor materials

DETAILED DESCRIPTION:
Thirty patients will be treated: 15 with a coronally positioned tunnel technique with NovaDerm® xenograft using continuous sling suture to secure both the graft and the flap (test treatment) and 15 with a coronally positioned tunnel technique with AlloDerm® allograft using continuous sling suture to secure both the graft and the flap (control treatment). Sutures used for the control group will be Maxon 5-0, 3/8 circle 13 mm needle for both the test and control groups. The coronally positioned tunnel technique was previously described by Edwards Pat Allen (E.P. Allen, Center for Advanced Dental Education, Dallas, Texas; course manual). Each patient will provide at least one Miller Class I or II facial recession defect, ≥ 3 mm. Patients will be randomly selected by a coin toss to receive either the test or control treatment. Mentor will toss the coin immediately prior to suturing. Patients will be evaluated postoperatively for a period of 4 months. The examiner will be blinded and will not be aware of the patient treatment at any time during the term of the study. Three exams for measurements will be performed per patient on total: preoperative, at week eight and 16 (4 months) postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* At least one Miller Class I or II mucogingival defect ≥ 3 mm (Miller 1985).
* The mucogingival defect must be on a non-molar tooth.
* Patients must be at least 18 years of age.

Exclusion Criteria:

* Patients with debilitating systemic or diseases that significantly affect the periodontium.
* Patients with a known allergy to any of the materials that will be used in the study, including systemic antibiotics (tetracycline and doxycycline).
* Patients requiring antibiotic prophylaxis.
* Root surface restorations at the site of recession.
* No detectable CEJ
* Patients who fail to maintain oral hygiene levels of at least 80% plaque free surfaces.
* Patients who are pregnant or lactating.
* Patients who use tobacco products (smoking or smokeless tobacco).
* Patients with alcohol abuse problems.
* Patients undergoing long-term steroid therapy.
* History of previous root coverage procedures, graft or GTR, on the test teeth.
* Patients who fail to complete the informed consent form.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-06 (Estimated); Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Percent root coverage | 4 months
  Initial and final recession will be measured from the cementoenamel junction to the gingival margin in millimeters. Root coverage will be determined by the amount of initial recession minus the final recession. Percent root coverage will be determined by root coverage divided by initial recession, multiplied by 100.

CONTACTS AND LOCATIONS:
Overall Officials: Henry Greenwell, DMD, MS, Principal Investigator — University of Louisville
Locations (1):
- Graduate Periodontics, UofL School of Dentistry, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No